CLINICAL TRIAL: NCT02299999
Title: PERSONALIZED MEDICINE GROUP / UCBG UC-0105/1304: SAFIR02_Breast - Evaluation of the Efficacy of High Throughput Genome Analysis as a Therapeutic Decision Tool for Patients With Metastatic Breast Cancer
Brief Title: SAFIR02_Breast - Efficacy of Genome Analysis as a Therapeutic Decision Tool for Patients With Metastatic Breast Cancer
Acronym: SAFIR02_Breast
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Fondation ARC (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0105/1304; 2013-001652-36 (EudraCT Number)
Record Dates: First submitted 2014-10-01; First posted 2014-11-24 (Estimated); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — vistusertib; AZD4547; capivasertib; AZD 8931; AZD 6244; vandetanib; bicalutamide; olaparib; Anthracyclines; Doxorubicin; Epirubicin; liposomal doxorubicin; Taxoids; Paclitaxel; Docetaxel; Cyclophosphamide; Methotrexate; Capecitabine; Fluorouracil; Gemcitabine; Vinca Alkaloids; Vinorelbine; Vinblastine; Vincristine; Platinum; Carboplatin; Cisplatin; Bevacizumab; Mitomycin; eribulin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Substudy 1: targeted agent (Experimental): Arm A1 / Targeted Arm : targeted maintenance from a list of 8 targeted drugs guided by the genomic analysis, AZD2014 tablet per os 50 mg bd, continuous dosing, AZD4547 tablet per os 80 mg bd, 2 weeks on/1 week off, AZD5363 capsule per os 480 mg bd, 4 days on/3 days off, AZD8931 tablet per os 40 mg bd, continuous dosing, selumetinib capsule per os 75 mg bd, continuous dosing, vandetanib tablet per os 300 mg od, continuous dosing, bicalutamide tablet per os 150 od, continuous dosing, olaparib tablet per os 300 mg bd, continuous dosing
  Interventions: Drug: AZD2014; Drug: AZD4547; Drug: AZD5363; Drug: AZD8931; Drug: Selumetinib; Drug: Vandetanib; Drug: Bicalutamide; Drug: Olaparib
- Substudy 1: standard maintenance therapy (Active Comparator): Arm B1/ maintenance Standard Chemotherapy Arm : such as Anthracyclines (Doxorubicin or Epirubicin or Liposomal Doxorubicine), Taxanes (Paclitaxel, Docetaxel), Cyclophosphamide, DNA Intercalators (Capecitabine, 5-FU, gemcitabine), Methotrexate, Vinca alkaloids (Vinorelbine, Vinblastine, Vincristine), Platinum based chemotherapies (Carboplatin, Cisplatin), Bevacizumab, Mitomycin C, Eribulin
  Interventions: Drug: Anthracyclines; Drug: Taxanes; Drug: cyclophosphamide; Drug: DNA intercalators; Drug: Methotrexate; Drug: vinca alkaloids; Drug: Platinum based chemotherapies; Drug: Bevacizumab; Drug: Mitomycin C; Drug: Eribulin
- Substudy 2: Immunotherapy (Experimental): Arm A2/ Immunotherapy arm: maintenance with MEDI4736 for patient without actionable genomic alterations or non eligible to Targeted substudy 1, MEDI4736 Intra-venous 10 mg/kg, Q2W
  Interventions: Drug: MEDI4736
- Substudy 2: standard maintenance therapy (Active Comparator): Arm B2/ maintenance Standard Chemotherapy Arm : such as Anthracyclines (Doxorubicin or Epirubicin or Liposomal Doxorubicine), Taxanes (Paclitaxel, Docetaxel), Cyclophosphamide, DNA Intercalators (Capecitabine, 5-FU, gemcitabine), Methotrexate, Vinca alkaloids (Vinorelbine, Vinblastine, Vincristine), Platinum based chemotherapies (Carboplatin, Cisplatin), Bevacizumab, Mitomycin C, Eribulin
  Interventions: Drug: Anthracyclines; Drug: Taxanes; Drug: cyclophosphamide; Drug: DNA intercalators; Drug: Methotrexate; Drug: vinca alkaloids; Drug: Platinum based chemotherapies; Drug: Bevacizumab; Drug: Mitomycin C; Drug: Eribulin

INTERVENTIONS:
Drug: AZD2014 — Target: m-TOR
  Arms: Substudy 1: targeted agent
Drug: AZD4547 — Target: EGFR
  Arms: Substudy 1: targeted agent
Drug: AZD5363 — Target: AKT
  Arms: Substudy 1: targeted agent
Drug: AZD8931 — Target: HER2, EGFR
  Arms: Substudy 1: targeted agent
Drug: Selumetinib — Target: MEK
  Other Names: ARRY-142866
  Arms: Substudy 1: targeted agent
Drug: Vandetanib — Target: VEGF, EGFR
  Other Names: CAPRELSA
  Arms: Substudy 1: targeted agent
Drug: Bicalutamide — target: Androgen receptor
  Other Names: Casodex
  Arms: Substudy 1: targeted agent
Drug: Olaparib — Target: PARP
  Other Names: Lynparza
  Arms: Substudy 1: targeted agent
Drug: Anthracyclines — DNA intercalation
  Other Names: Doxorubicin, Epirubicin, liposomal doxorubicin
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: Taxanes — Target: mitotic tubulin and microtubules
  Other Names: paclitaxel; docetaxel
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: cyclophosphamide — Alkylating agents
  Other Names: Novatrex; Imeth
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: DNA intercalators — DNA intercalators
  Other Names: capecitabine; 5-FU; gemcitabine
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: Methotrexate — DNA intercalators
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: vinca alkaloids — Target: mitotic tubulin and microtubules
  Other Names: vinorelbine; vinblastine; vincristine
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: Platinum based chemotherapies — Platinum based chemotherapies
  Other Names: Platinum; carboplatin; cisplatin
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: Bevacizumab — Target: VEGF
  Other Names: Avastin
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: Mitomycin C — Alkylating agents
  Other Names: Ametycine
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: Eribulin — Microtubule modulator
  Other Names: Halaven
  Arms: Substudy 1: standard maintenance therapy; Substudy 2: standard maintenance therapy
Drug: MEDI4736 — Target: PD-L1
  Arms: Substudy 2: Immunotherapy

SUMMARY:
Open label multicentric phase II randomized trial, using high throughput genome analysis as a therapeutic decision tool, which aims at comparing a targeted treatment administered according to the identified molecular anomalies of the tumor with maintenance chemotherapy (targeted substudy 1) as well as immunotherapy with maintenance chemotherapy in patients without actionable genomic alterations or non eligible to substudy 1 (immune substudy 2).

DETAILED DESCRIPTION:
Screening phase:

New frozen biopsy or an archived frozen sample or ctDNA sample will be sent to the genomic platforms for DNA extraction and genomic analysis (DNA microarrays and Next generation sequencing).

Patients can be considered as pre-eligible for the targeted substudy 1 randomisation phase when both following mandatory conditions have been met: stable or responding disease has been observed (investigator judgment) after 6 to 8 cycles of chemotherapy (or at least after 4 cycles of chemotherapy if stopped for toxicity) and targetable alteration has been identified by the Molecular Tumor Board (MTB).

If not eligible for the substudy 1 randomisation phase, patients can be considered as pre-eligible for the immune substudy 2 randomization phase when both following mandatory conditions are met: stable or responding disease (investigator judgment) is observed after 6 to 8 cycles of chemotherapy (or at least after 4 cycles if treatment was stopped due to toxicity) AND not eligible to randomization in the substudy 1 (because patient had no targetable alteration identified by the Molecular Tumor Board, or failed to have a genomic profile for the tumor [low tumor cells percentage, technical issue during genomic analysis, etc.], or a non inclusion criteria that precluded entry into the substudy 1)

Randomization phase:

The mandatory post-chemotherapy wash-out period, of 28 days for 21 or 28 day-cycle chemotherapies or of 15 days for weekly (except monoclonal antibodies) or daily chemotherapies,will provide time to achieve all the required tests and examinations.

The randomization program will allocate the following treatments with a 2:1 ratio in favor of Arm A of the considered substudy:

Substudy 1 : targeted therapies versus standard maintenance chemotherapy

* Arm A1 / targeted arm: targeted maintenance from a list of 8 targeted drugs guided by the genomic analysis, or
* Arm B1 / chemotherapy arm : maintenance chemotherapy (or no antineoplastic treatment in case of toxicity at the time of randomization)

Substudy 2 : immunotherapy versus standard maintenance chemotherapy

* Arm A2 / immunotherapy maintenance arm: MEDI4736 or
* Arm B2 / chemotherapy arm: chemotherapy continued as a maintenance chemotherapy (or no antineoplastic treatment in case of toxicity)

ELIGIBILITY:
Screening phase:

Inclusion Criteria:

* Women (or men) with histologically proven breast cancer
* Metastatic relapse or progression or stage IV at diagnosis
* No Her2 over-expression
* Patients with metastases that can be biopsied, except bone metastases
* Patients who are eligible for a first or a second line of chemotherapy in metastatic setting (left to the discretion of investigators), or who are currently treated with a first or second line of chemotherapy with a maximum of 2 cycles at the time of biopsy. Screening of patients currently treated with a second line chemotherapy should have a stable disease
* For patients with ER+ disease, relapse or progression occurred during endocrine therapy, whatever the line, or less than 12 months after the end of endocrine therapy in adjuvant context
* Age ≥18 years
* WHO Performance Status 0/1
* Presence of measurable target lesion according to RECIST criteria v1.1

Exclusion criteria:

* Spinal cord compression and/or symptomatic or progressive brain metastases
* Bone metastases when this is the only site of biopsiable disease
* Patients with all target lesions in a previously irradiated region, except if clear progression has been observed prior to study in at least one of them
* Patient who received more than 2 lines of chemotherapy at the time of the biopsy
* Tumor progression observed with the current line of treatment when under 2nd line
* Patients who already had a genomic profile (both CGH and NGS analysis) in which no SAFIR02 targetable alterations have been identified
* Abnormal coagulation contraindicating biopsy
* Inability to swallow
* Major problem with intestinal absorption Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG Any factors increasing the risk of QTc prolongation or arrhythmic events Experience of any of the following in the preceding 12 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, past or current uncontrolled angina pectoris, congestive heart failure NYHA Grade ≥2, torsades de pointes, current uncontrolled hypertension, cardiomyopathy Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which requires steroid treatment or any evidence of clinically interstitial lung disease Previous or current malignancies of other histologies within the last 5 years, Evidence of severe or uncontrolled systemic disease (active bleeding diatheses, or active Hepatitis B, C and HIV)
* diagnosis of acne rosacea, severe psoriasis and severe atopic eczema
* Prior exposure to anthracyclines or mitoxantrone with cumulative exposure in excess of 360 mg/m² for doxorubicin, 720 mg/m² for epirubicin, or 72 mg/m² for mitoxantrone
* Previous treatment with the same agent or in the same class as one of those used in the SAFIR02 trial (patients who received this previous targeted agent without the target prescreening are eligible but may not be eligible for randomisation in substudy 1 if the treatment allocated by the MTB is in the same class) History of retinal degenerative disease, eye injury or corneal surgery in the previous 3 months, past history of central serous retinopathy or retinal vein occlusion, intraocular pressure >21 mmHg, or uncontrolled glaucoma.
* History of hemorrhagic or thrombotic stroke, TIA or other CNS bleeds
* Renal disease including glomerulonephritis, nephritic syndrome, Fanconi syndrome, renal tubular acidosis
* Patients using drugs that are known potent inhibitors or potent inducers or substrates of cytochrome P450

Randomized phase:

Substudy 1:

Inclusion Criteria:

* Patients who received 6 to 8 cycles of chemotherapy, or having received at least 4 cycles of chemotherapy definitively stopped for toxicity reasons, and who are presenting a SD or PR at randomization
* presenting at least one genomic alteration from the predefined list
* Age ≥25 years for patients planned to receive AZD4547
* 28-day wash-out period from chemo prior to randomization and grade ≤1 residual toxicities

Exclusion Criteria:

* More than 2 previous lines of chemotherapy for metastatic disease before randomization
* Life expectancy <3 months
* Disease progression occuring at any time during chemotherapy and before randomization or toxicity that led to the discontinuation of the last chemotherapy before 4 full cycles have been delivered
* Less than 28 days from radiotherapy, less than 2 weeks from palliative radiation
* Patients previously treated with a targeted agent in the same class as the agent to be given to the patient in substudy 1
* Toxicities of grade ≥2 from any previous anti-cancer therapy
* Altered haematopoietic or organ function
* Mean resting corrected QT interval (QTc) >480 msec (or QTcF >450 msec) obtained from 3 consecutive ECGs
* Left ventricular ejection fraction (LVEF) <55% (MUGA scan or Echocardiogram)
* Altered ophthalmic conditions confirmed by an ophthalmology specialist for patients likely to be treated with AZD4547 orAZD8931 or Selumetinib
* Patients using non-substitutable drugs, that are known to prolong QT interval or induce Torsades de Pointes, when they are supposed to be treated with vandetanib, AZD5363 or AZD8931

Substudy 2:

Inclusion Criteria:

* Patients who received 6 to 8 cycles of chemotherapy, or having received at least 4 cycles of chemotherapy definitively stopped for toxicity reasons, and who are presenting a SD or a RP at randomization
* Patients not eligible to substudy 1
* wash-out period of at least 15 days for weekly (except monoclonal antibodies) or daily chemotherapies or 28 days for other chemotherapies from last chemotherapy administration prior to randomization and grade ≤1 residual toxicities

Exclusion Criteria:

* More than 2 previous lines of chemotherapy for metastatic disease before randomization
* Life expectancy <3 months
* Disease progression occuring at any time during chemotherapy and before randomization or toxicity that led to the discontinuation of the last chemotherapy before 4 full cycles have been delivered
* Any previous treatment with a PD1 or PD-L1 inhibitor, including MEDI4736
* Toxicities of grade ≥2 from any previous anti-cancer therapy
* Altered haematopoietic or organ function
* Mean resting QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 consecutive ECGs using Bazett's Correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of MEDI4736, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* History of primary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1460 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival in the targeted drug arm compared to standard maintenance therapy arm | from randomization to disease progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  To evaluate whether treatment with targeted agents guided by high throughput molecular analysis (CGH array, next generation sequencing) improves progression-free survival as compared to standard maintenance therapy in patients with metastatic Breast Cancer

SECONDARY OUTCOMES:
progression-free survival in patients treated with anti-PDL1 antibody (MEDI4736) compared to standard maintenance therapy arm | from randomization to disease progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  To evaluate whether treatment with MEDI4736 improves progression-free survival as compared to standard maintenance therapy in patients with metastatic Breast Cancer
overall survival in each substudy | from randomization to death (any cause), up to 16 months
  To evaluate whether treatment with targeted agents guided by high throughput molecular analysis (CGH array, next generation sequencing) or MEDI4736 improves overall survival as compared to standard maintenance therapy in patients with metastatic Breast Cancer
overall response rates and changes in tumor size in each substudy | tumor response is assessed every 21 days from treatment initiation until first progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  tumor response is defined as a complete or partial response, upon RECIST v1.1 criteria
evaluate safety, in each substudy | toxicities will be assessed during the whole treatment period (4 months expected in average) followed by a 1-year post-treatment follow-up period, and reported during the visits scheduled by the study flow chart
  Toxicities are graded according to the CTCAE V4
efficacy (response rate, change in tumor size, progression-free survival, overall survival) and safety of each individual targeted agent (substudy 1) | tumor response is assessed every 21 days from treatment initiation until first progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  tumor response is defined as a complete or partial response, upon RECIST v1.1 criteria
correlate molecular characteristics in patients with the efficacy endpoints (response rate, progression-free and overall survival) in each substudy | from randomization or treatment initiation to disease progression or death from any cause, whichever comes first, up to 16 months (estimated treatment duration average: 4 months)
  tumor response is defined as a complete or partial response, upon RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice ANDRE, Pr, Principal Investigator — Gustave Roussy, Villejuif
Locations (25):
- France (25):
  - Institut de Cancérologie de l'Ouest/Paul Papin, Angers
  - Institut Sainte-Catherine, Avignon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Chd Vendee, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Chu Dupuytren, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Régional du Cancer Montpellier Val d'Aurelle, Montpellier
  - Centre Alexis Vautrin, Nancy
  - Institut de Cancérologie de l'Ouest/ René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie, Saint-Cloud
  - Hopitaux Universitaire de Strasbourg - Hopital Civil, Strasbourg
  - Hopitaux Du Leman, Thonon-les-Bains
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mosele F, Stefanovska B, Lusque A, Tran Dien A, Garberis I, Droin N, Le Tourneau C, Sablin MP, Lacroix L, Enrico D, Miran I, Jovelet C, Bieche I, Soria JC, Bertucci F, Bonnefoi H, Campone M, Dalenc F, Bachelot T, Jacquet A, Jimenez M, Andre F. Outcome and molecular landscape of patients with PIK3CA-mutated metastatic breast cancer. Ann Oncol. 2020 Mar;31(3):377-386. doi: 10.1016/j.annonc.2019.11.006. Epub 2020 Jan 24. PMID 32067679
- See also: Unicancer official website — http://www.unicancer.fr/
- See also: SAFIR01 study results — http://www.ncbi.nlm.nih.gov/pubmed/24508104